CLINICAL TRIAL: NCT01764048
Title: To Compare the Efficacy and Patient's Satisfaction From Pain Management of Women After Cesarean Section by Pain Relievers' Administration in Fix Protocol Compared to Protocol Following Demand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0120-12-EMC
Record Dates: First submitted 2013-01-02; First posted 2013-01-09 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Pain Management; Cesarean Section
Keywords: pain management; cesarean section
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fix protocol (Experimental): During 48 hours following surgery pain medications will be given as followed (listed in brackets are the generic names of each medication):
  At patient arrival to the department: Intravenous Tramadol hydrochloride 100 milligrams + TAB. Paracetamol 500 milligrams + TAB. Diclofenac 100 milligrams
  After 6 hours from patient arrival and every 6 hours: TAB. Zaldiar (Paracetamol 650 milligrams + Tramadol 75 milligrams).
  After 12, 24 and 48 hours from patient arrival: TAB. Diclofenac 100 milligrams.
  Rescue medication: TAB. Percocet (Oxycodone 5MG/Paracetamol 325 MG)as necessary up to 4 times per day.
  The total amount of paracetamol is limited to 4 gr per day.
  Interventions: Drug: Fix protocol
- medications following demand protocol (Experimental): The same combinations will be given as in the fixed protocol however only after patient request
  Interventions: Drug: medications following demand protocol

INTERVENTIONS:
Drug: Fix protocol — Please see arm description
  Arms: Fix protocol
Drug: medications following demand protocol — Please see arm description
  Arms: medications following demand protocol

SUMMARY:
Cesarean deliveries are prevalent. Unlike other operations, quick recovery is required for the mother to nurture the newborn child and establishing an appropriate mother-child bonding. Therefore, effective pain management is crucial. In this study we would like to compare between two pain relievers' administration protocols: (1) pain relievers' administration in fix protocol (type of medications, dose and intervals) or (2) pain relievers' administration following demand (the same type and doses, however, medications will be given only following patient's request).

The primary outcome will be patient satisfaction, pain control and the necessity of additional medications (rescue doses).

The protocols will be used for the first 48 hours following surgery.

ELIGIBILITY:
Inclusion Criteria:

* women that underwent cesarean section

Exclusion Criteria:

* Women suffering from chronic pain
* Women using chronic pain medications
* Allergy to any drug used in the study
* Women underwent general anesthesia during the surgery
* women with elevated liver enzymes

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 214 (Actual)
Dates: Start 2012-11; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The efficacy of pain management | during 48 hours from surgery
  Pain sensation will be assessed using the VAS scale (visual analog scale) for measurement of acute pain

SECONDARY OUTCOMES:
adverse effect of the medications given in each protocol | during 48 hours following surgery
to compare the amount of breastfeeding between 2 groups | following the week after surgery
The number of times that pain medications were given in each study group | during 48 hours following surgery
The necessity of additional medications (rescue doses) | During 48 hours after surgery
Patient satisfaction | 48 hours after surgery
  Each patient will fill in a satisfaction questioner which is given 48 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of obstetric and gynecology, HaEmek medical center, Afula, Israel